CLINICAL TRIAL: NCT02657161
Title: Phase I Study to Determine the Safety and Efficacy of a PIKA Rabies Vaccine Containing the PIKA Adjuvant
Brief Title: Safety and Efficacy of a PIKA Rabies Vaccine Containing the PIKA Adjuvant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yisheng Biopharma (Singapore) Pte. Ltd. (Industry)
Collaborators: Duke-NUS Graduate Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RV001-I
Record Dates: First submitted 2016-01-11; First posted 2016-01-15 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Rabies
MeSH Terms: conditions — Rabies | interventions — PIKA adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A (Active Comparator): Comparator vaccine RABIPUR®
  Healthy volunteers received rabies vaccination intramuscularly on days 0,3,7 and 14
  Interventions: Biological: RABIPUR®
- Group B (Experimental): PIKA Rabies vaccine
  Healthy volunteers received rabies vaccination intramuscularly on days 0,3,7 and 14
  Interventions: Biological: PIKA rabies vaccine
- Group C (Experimental): PIKA Rabies vaccine with an accelerated regimen
  Healthy volunteers received rabies vaccination intramuscularly on days 0 (2 Doses), 3 (2 Doses), and day 7 (1 Dose)
  Interventions: Biological: PIKA rabies vaccine with an accelerated regimen

INTERVENTIONS:
Biological: RABIPUR® — Biological rabies vaccine
  Arms: Group A
Biological: PIKA rabies vaccine — Biological rabies vaccine
  Other Names: 'PIKA rabies vaccine with PIKA adjuvant
  Arms: Group B
Biological: PIKA rabies vaccine with an accelerated regimen — Biological rabies vaccine
  Other Names: 'PIKA rabies vaccine with PIKA adjuvant
  Arms: Group C

SUMMARY:
Phase I clinical study for an investigational PIKA (Polyinosinic-Polycytidylic Acid Based Adjuvant) rabies vaccine comprising Inactivated and Purified Rabies Virus (IPRV) and the PIKA adjuvant. The primary objective of the study was to assess the clinical safety of the vaccine composition in healthy adult volunteers. The secondary objective was to evaluate the vaccine's efficacy based on an accelerated vaccine regimen.

DETAILED DESCRIPTION:
A single-center, open label, randomized phase I study in healthy naïve adult subjects. There were three study groups; subjects were randomly assigned to groups A (12), B (12) and C (12). Group A, as a control arm of the study, had received a commercially available rabies vaccine, RABIPUR® and Group B had received doses of the investigational PIKA rabies vaccine. Group C received an accelerated vaccine regimen with the investigational PIKA rabies vaccine. Group A and B followed the same vaccine regimen of (1-1-1-1), one injection on days 0, 3, 7 and 14 was administered respectively. Group C received the accelerated regimen (2-2-1), two injections on both days 0 and 3 were administered in different arms; and only one injection was administered on day 7.

Each vaccine dose comprise 1.0 ml of PIKA rabies vaccine for Group B and Group C and 1.0 ml of RABIPUR® for Group A after reconstitution. The route of administration is intramuscular injection, given in the deltoid region of the arm.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent form has been signed and dated
* Able to attend all scheduled visits and comply with all trial procedures.
* Never received rabies vaccine before.
* Refrain from blood donation during the course of the study.
* Able to attend all scheduled visits and comply with all trial procedures.

Exclusion Criteria:

* For women who are pregnant and breast-feeding
* Previous vaccination against rabies (in pre- or post-exposure regimen) with either the trial vaccine or another vaccine
* History of allergies to the medicine (S), convulsions, epilepsy, mental illness and brain disease and clear serious systemic reaction
* Known bleeding disorder or suspected impairment of immunologic function, or receipt of immunosuppressive therapy or immunoglobulin since birth
* Participation in any other interventional clinical trial
* Donation of blood within the last 2 months or who have donated plasma within the last 14 days
* Patient with clinical signs of encephalitis
* Recipient of any vaccine in the 4 weeks preceding the first trial vaccination, except for influenza vaccination
* Concomitant use or at high probability of expected concomitant use during the planned study of medication such as immune suppressants, steroids, non-study vaccine or similar substances
* Use of any investigational or non-registered drug or vaccine other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Administration of immunoglobulins and/or any blood products within 3 months prior to the first dose of study vaccine or planned administration during the study period.
* History of allergic disease or reactions likely to be exacerbated by any component of the study vaccines.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* Uncontrolled acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by medical history or physical examination.
* Chronic administration of immuno-suppressants or other immune-modifying drugs within 3 months prior to the first vaccine dose.
* Clinical Manifestation of Metabolic, blood system, lungs, heart, the gastrointestinal tract, nervous system, kidneys, urinary system, endocrine, liver disease or malignant tumor

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2015-02; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Identification of any adverse events for all the treatment groups | 42 days
  Assessment of safety based on the identification of any adverse events for all the treatment groups, Group A, Group B and Group C through to the end of the study at day 42.
Titer level of Rabies Virus Neutralizing Antibody (RVNA) from serum at day 14 and 42 after the first injection | Day 14 and Day 42
  To analyze the titer level of RVNA from serum at day 14 and 42 after the first injection and with RVNA titer meeting the 0.5 IU(International units) /ml World Health Organization (WHO) requirement

SECONDARY OUTCOMES:
Detectable specific T cell mediated immune response on day 7 or day 14 and 42 | Day 7, Day 14 and Day 42
  Assessment of efficacy was determined by the observed immune response in subjects receiving the investigational vaccine where:Detectable specific T cell mediated immune response on day 7 or day 14 and 42
Number of subjects in Group C who has higher RVNA titre level on Day 7 or Day 14 when compared to classic course. | Day 7 and Day 14
  Evaluation of the accelerated regimen is studied to check if the levels of anti-rabies antibodies (serum RVNA titer) will be higher in day 7 or 14 than a classic course with control commercialized vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: Limin Wijaya, Principal Investigator — Singapore General Hospital
Locations (1):
- SingHealth Investigational Medicine Unit, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yu P, Liu Y, Tao X, He Y, Liu Q, Wang B, Zheng H, Zhang N, Bi S, Zhu W, Zhang Y. Potential option for rabies post-exposure prophylaxis: New vaccine with PIKA adjuvant against diverse Chinese rabies strains. Vaccine. 2023 Nov 2;41(46):6852-6862. doi: 10.1016/j.vaccine.2023.10.001. Epub 2023 Oct 9. PMID 37821317
- [Derived] Wijaya L, Tham CYL, Chan YFZ, Wong AWL, Li LT, Wang LF, Bertoletti A, Low JG. An accelerated rabies vaccine schedule based on toll-like receptor 3 (TLR3) agonist PIKA adjuvant augments rabies virus specific antibody and T cell response in healthy adult volunteers. Vaccine. 2017 Feb 22;35(8):1175-1183. doi: 10.1016/j.vaccine.2016.12.031. Epub 2017 Jan 22. PMID 28118938